CLINICAL TRIAL: NCT04411238
Title: Skills of Home Helpers for a Better Quality of Life for Adults With Huntington's Disease Living at Home
Acronym: COMPQUAHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/28
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Quality of Life
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients
  Interventions: Other: interview
- Caregivers
  Interventions: Other: interview
- Home help
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — interview

SUMMARY:
Huntington's disease often brings together 3 types of symptoms at one time or another of the disease during its evolution: motor, cognitive and psychiatric. Management requires comprehensive and multidisciplinary health, social or medico-social support. Its development generates additional difficulties for professionals who very often qualify this disease as "very complex" because it leads to a deep and severe impairment of physical and intellectual capacities. The sick person gradually loses their autonomy and becomes dependent for the acts of daily life, hence the choice of this disease for our study. Our study is focused on the quality of life at home of patients followed by the Angers Reference Center, "expert" on neurogenetic pathologies.

Studies focusing on patients' quality of life at home have so far never been undertaken for a rare neurodegenerative disease like Huntington's disease.

ELIGIBILITY:
Selection Criteria:

Patient group :

* Genetic diagnosis of Huntington's disease
* Symptomatic patient
* Patient living at home
* Person able to carry out the interviews provided for in the study

Caregiver group :

* Person, defined within the meaning of the CNSA (National Solidarity Fund for Autonomy) as a natural caregiver, not concerned himself by the risk of developing the disease
* person able to carry out the interviews provided for in the study

Home Helper group :

- Professionals working at home with Huntington's disease patients employed by home help service providers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 90 participants, including 30 cases with Huntington's disease, 30 caregivers not concerned himself with the risk of developing the disease and 30 home helper worker for Huntington's disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Identify and compare the expectations and needs of patients with Huntington's disease, their caregivers, and home helpers, in terms of home support, based on interviews | One day